CLINICAL TRIAL: NCT00434785
Title: An Ascending, Multiple Dose Study of the Safety, Tolerability, and Pharmacokinetics of AGG-523 Administered Orally to Healthy Male Japanese Subjects.
Brief Title: A Study of the Safety, Tolerability, and Pharmacokinetics of AGG-523 in Healthy Japanese Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3189A1-105
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Healthy

INTERVENTIONS:
Drug: AGG-523

SUMMARY:
To assess the safety and tolerability of ascending, multiple oral doses of AGG-523 in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 20 to 40 years, inclusive, at screening; sexually active men must agree to use a medically acceptable form of contraception during the study and continue for 12 weeks after test article administration.
* Body mass index (BMI) in the range of 17.6 to 26.4 Kgm2, and body weight >45 kg.
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12 lead ECG.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-02; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To assess the safety and PK profile

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Ikebukuro, Tokyo, Japan